CLINICAL TRIAL: NCT00210470
Title: A Phase 2, Open-label Trial of the Safety and Biological Effect of Subcutaneous IRX-2 (With Cyclophosphamide, Indomethacin, and Zinc) in Patients With Resectable Cancer of the Head and Neck
Brief Title: A Phase 2 Clinical Trial of the Safety and Effects of IRX-2 in Treating Patients With Operable Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brooklyn ImmunoTherapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRX-2 2005-A
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-02-08 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and Neck Cancer; Immunotherapy; IRX-2; Mouth Cancer; Throat Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Mouth Neoplasms | interventions — IRX 2; Cyclophosphamide; Indomethacin; Zinc; gluconic acid; Omeprazole

STUDY DESIGN:
Intervention Model Description: Open Label Single Arm Phase 2a trial of Safety of IRX-2 in Patients with Operable Head and Neck Cancer
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IRX-2 Regimen (Experimental): The IRX-2 regimen is the combination of a 2-week course of IRX-2 itself, an initial dose of cyclophosphamide, and a 3-week course of indomethacin, zinc supplementation, and omeprazole.
  Interventions: Biological: IRX-2; Drug: Cyclophosphamide; Drug: Indomethacin; Drug: Zinc; Drug: Omeprazole

INTERVENTIONS:
Biological: IRX-2 — IRX-2 for 10 days (2 s.c. injections of 1 mL each day) into bilateral mastoid insertion regions.
Drug: Cyclophosphamide — Single i.v. injection of low-dose (300 mg/m2) on Day 1
  Other Names: Cytoxan; cyclophosphane
Drug: Indomethacin — 21 days of oral indomethacin, 25 mg. 3 times daily
  Other Names: Indocin; Indocid
Drug: Zinc — 21 days of zinc gluconate (65 mg) as part of an oral multivitamin
  Other Names: zinc gluconate
Drug: Omeprazole — 21 days of 20 mg. orally
  Other Names: Prilosec

SUMMARY:
This was a Phase 2a trial to investigate the safety and biological activity of the RIX-2 Regimen in patients with untreated, resectable squamous cell cancer of the head and neck (HNSCC).

DETAILED DESCRIPTION:
IRX-2 is a primary cell-derived biologic that reduces the immune suppression that is often seen in the cancer tumor micro-environment, restores immune function and activates a coordinated immune response against the tumor. IRX-2 is a complex proprietary therapeutic containing numerous active cytokine components, which restores and activates multiple immune cell types including T cells, dendritic cells, and natural killer cells to recognize and destroy tumors.

The present study administered the IRX-2 Regimen to 27 patients as a neoadjuvant (before surgery) therapy, and the main objective of the study was to determine the safety and tolerability of the IRX-2 regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed (histology) Squamous Cell Carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx.
* No prior surgery, radiation therapy or chemotherapy of this tumor other than biopsy or emergency procedure required for supportive care.
* Clinically staged Stage II, III, or IVA cancer, assessed to be surgically resectable with curative intent.
* Life Expectancy of greater than 6 months

Exclusion Criteria:

* Stage IVB Squamous Cell Carcinoma
* Use of any investigational agent within the previous 30 days
* Uncontrolled cardiovascular disease
* Myocardial infarction within the last 3 months
* Abnormal hemoglobin, neutrophil, lymphocyte or platelet counts
* Positive for hepatitis B or C or HIV
* Evidence of distant metastases
* Clinical gastritis or peptic ulcer within the last 6 months
* Stroke within the last six months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-07; Primary Completion 2010-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Moyer, MD, Principal Investigator — University of Michigan Hospitals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schilling B, Harasymczuk M, Schuler P, Egan JE, Whiteside TL. IRX-2, a novel biologic, favors the expansion of T effector over T regulatory cells in a human tumor microenvironment model. J Mol Med (Berl). 2012 Feb;90(2):139-47. doi: 10.1007/s00109-011-0813-8. Epub 2011 Sep 14. PMID 21915712
- [Background] Czystowska M, Szczepanski MJ, Szajnik M, Quadrini K, Brandwein H, Hadden JW, Whiteside TL. Mechanisms of T-cell protection from death by IRX-2: a new immunotherapeutic. Cancer Immunol Immunother. 2011 Apr;60(4):495-506. doi: 10.1007/s00262-010-0951-9. Epub 2010 Dec 23. PMID 21181158
- [Background] Naylor PH, Hernandez KE, Nixon AE, Brandwein HJ, Haas GP, Wang CY, Hadden JW. IRX-2 increases the T cell-specific immune response to protein/peptide vaccines. Vaccine. 2010 Oct 8;28(43):7054-62. doi: 10.1016/j.vaccine.2010.08.014. Epub 2010 Aug 13. PMID 20708999
- [Background] Naylor PH, Hadden JW. Preclinical studies with IRX-2 and thymosin alpha1 in combination therapy. Ann N Y Acad Sci. 2010 Apr;1194:162-8. doi: 10.1111/j.1749-6632.2010.05475.x. PMID 20536465
- [Background] Rapidis AD, Wolf GT. Immunotherapy of head and neck cancer: current and future considerations. J Oncol. 2009;2009:346345. doi: 10.1155/2009/346345. Epub 2009 Aug 9. PMID 19680453
- [Background] Czystowska M, Han J, Szczepanski MJ, Szajnik M, Quadrini K, Brandwein H, Hadden JW, Signorelli K, Whiteside TL. IRX-2, a novel immunotherapeutic, protects human T cells from tumor-induced cell death. Cell Death Differ. 2009 May;16(5):708-18. doi: 10.1038/cdd.2008.197. Epub 2009 Jan 30. PMID 19180118
- [Background] Bright J, Al-Shamahi A. BioPartnering Europe--15th Annual Conference. Highlights from open house and emerging company presentations--Part 1. IDrugs. 2007 Dec;10(12):855-7. No abstract available. PMID 18041679
- [Background] Egan JE, Quadrini KJ, Santiago-Schwarz F, Hadden JW, Brandwein HJ, Signorelli KL. IRX-2, a novel in vivo immunotherapeutic, induces maturation and activation of human dendritic cells in vitro. J Immunother. 2007 Sep;30(6):624-33. doi: 10.1097/CJI.0b013e3180691593. PMID 17667526
- [Background] Hadden JW, Verastegui E, Hadden E. IRX-2 and thymosin alpha1 (Zadaxin) increase T lymphocytes in T lymphocytopenic mice and humans. Ann N Y Acad Sci. 2007 Sep;1112:245-55. doi: 10.1196/annals.1415.032. Epub 2007 Jun 28. PMID 17600288
- [Background] Naylor PH, Quadrini K, Garaci E, Rasi G, Hadden JW. Immunopharmacology of thymosin alpha1 and cytokine synergy. Ann N Y Acad Sci. 2007 Sep;1112:235-44. doi: 10.1196/annals.1415.036. Epub 2007 Jun 13. PMID 17567942
- [Background] Bayes M, Rabasseda X, Prous JR. Gateways to clinical trials. Methods Find Exp Clin Pharmacol. 2004 Sep;26(7):587-612. PMID 15538546
- [Background] Hadden JW. Immunodeficiency and cancer: prospects for correction. Int Immunopharmacol. 2003 Aug;3(8):1061-71. doi: 10.1016/S1567-5769(03)00060-2. PMID 12860163
- [Result] Freeman SM, Franco JL, Kenady DE, Baltzer L, Roth Z, Brandwein HJ, Hadden JW. A phase 1 safety study of an IRX-2 regimen in patients with squamous cell carcinoma of the head and neck. Am J Clin Oncol. 2011 Apr;34(2):173-8. doi: 10.1097/COC.0b013e3181dbb9d8. PMID 20539208
- [Result] Wolf GT, Fee WE Jr, Dolan RW, Moyer JS, Kaplan MJ, Spring PM, Suen J, Kenady DE, Newman JG, Carroll WR, Gillespie MB, Freeman SM, Baltzer L, Kirkley TD, Brandwein HJ, Hadden JW. Novel neoadjuvant immunotherapy regimen safety and survival in head and neck squamous cell cancer. Head Neck. 2011 Dec;33(12):1666-74. doi: 10.1002/hed.21660. Epub 2011 Jan 31. PMID 21284052
- [Result] Berinstein NL, Wolf GT, Naylor PH, Baltzer L, Egan JE, Brandwein HJ, Whiteside TL, Goldstein LC, El-Naggar A, Badoual C, Fridman WH, White JM, Hadden JW. Increased lymphocyte infiltration in patients with head and neck cancer treated with the IRX-2 immunotherapy regimen. Cancer Immunol Immunother. 2012 Jun;61(6):771-82. doi: 10.1007/s00262-011-1134-z. Epub 2011 Nov 6. PMID 22057678
- [Result] Whiteside TL, Butterfield LH, Naylor PH, Egan JE, Hadden JW, Baltzer L, Wolf GT, Berinstein NL. A short course of neoadjuvant IRX-2 induces changes in peripheral blood lymphocyte subsets of patients with head and neck squamous cell carcinoma. Cancer Immunol Immunother. 2012 Jun;61(6):783-8. doi: 10.1007/s00262-011-1136-x. Epub 2011 Nov 23. PMID 22109700
- See also: IRX Therapeutics website — http://www.irxtherapeutics.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled July 2005 and the last subject visit was August 2009.
Pre-assignment Details: Pathologically confirmed (by histology) squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx.
  No prior surgery, radiation therapy, or chemotherapy of this tumor other than biopsy or emergency procedure required for supportive care.
  No medical contraindications to surgical resection and reconstruction required.
Groups:
- IRX-2 Regimen: The IRX-2 regimen is the combination of a 2-week course of IRX-2 itself, an initial dose of cyclophosphamide, and a 3-week course of indomethacin and zinc supplementation.
Period: Overall Study
Arm/Group | IRX-2 Regimen
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 26
  Mexico | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: The frequency of all Adverse Events (greater than 5%) is reported. All Serious Adverse Events were described.
Time Frame: Enrollment through 30 days post-surgery
Population: 27 participants were entered into study and treated. All participants were included in the safety analysis.
Measure: Count of Participants; unit: Participants
Groups:
- IRX-2 Regimen: A 2-week course of IRX-2, an initial low dose of cyclophosphamide, and a 3-week course of indomethacin and zinc supplementation
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 27
Participants
  Adverse Event: Injection Site Pain | 6
  Adverse Event: Headache | 8
  Adverse Event: Nausea | 6
  Adverse Event: Constipation | 4
  Adverse Event: Dizziness | 4
  Adverse Event: Fatigue | 3
  Adverse Event: Pneumonia Aspiration | 3
  Adverse Event: Anaemia | 3
  Adverse Event: Injection Site Discomfort | 3
  Adverse Event: Myalgia | 2
  Adverse Event: Contusion | 2
  Adverse Event: Dry Mouth | 2
  Adverse Event: Vomiting | 2
  Additional AE Categories w lower frequency | 4
  Serious Adverse Events | 7

2. Secondary Outcome: Clinical and Histological Tumor Responses
Description: Number of participants with the specified percent change in size of target lesion is presented
Time Frame: On approximately Day 21 (last day of treatment) prior to undergoing post-treatment surgery
Population: A total of 23 subjects who received the IRX-2 regimen were evaluated for tumor response based on the RECIST criteria
Measure: Count of Participants; unit: Participants
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 23
Participants
  -20% to < -10% | 4
  -10% to < 0% | 7
  0% to < 10% | 9
  10% to < 20% | 1
  20% to < 30% | 0
  >= 30% | 2
Statistical Analysis 1: Comparison: IRX-2 Regimen; Test type: Equivalence — The correlation of each of the above variables at biopsy/Day 1, surgery/Day 21, and change with percent change in the longest diameter (LD) of the primary tumor was calculated using Spearman rank correlations (183 correlations). Due to outliers in the distribution of percent change in the longest diameter, it was felt that the Spearman rank correlations would be more appropriate than Pearson correlations; p < 0.10, Spearman Rank

3. Secondary Outcome: Patient Tolerance of Surgery and Post-operative Adjuvant Therapy;
Description: Patient Tolerance of Surgery and Post-operative Adjuvant Therapy as measured by median days spent in the hospital, intensive care unit, and step down unit.
Time Frame: Following surgery and post-operative therapy (up to 39 days post surgery)
Population: Following surgery the median days spent in the hospital, intensive care unit and step down unit was determined for 26 subjects
Measure: Median (Full Range); unit: days
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 26
days
  Median Days in hospital | 8.5 [1 to 39]
  Median Days in intensive care unit | 0.5 [0 to 17]
  Median Days in step-down unit | 0.5 [0 to 22]

4. Secondary Outcome: Immune Competence as Measured by Skin Test Reactivity
Description: To assess measures of immune competence following administration of the IRX-2 regimen, including skin test reactivity.
Time Frame: At approx. 21 days, prior to surgery
Population: Skin response (erythema) was evaluated at Baseline and Day 21 on 26 subjects treated with IRX-2 Regimen
Measure: Count of Participants; unit: Participants
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 26
Participants
  Positive at both Baseline and at Day 21 (%) | 12
  Negative at both Baseline and Day 21 (%) | 6
  Positive at Baseline and Negative Day 21 (%) | 6
  Negative at Baseline and Positive at Day 21 | 2
  Induration at Day 21 | 3

5. Secondary Outcome: Disease-free Survival
Description: Estimate disease-free survival (DFS) (time from surgery to death or clinically apparent, biopsy confirmed recurrent or progressive disease after the completion of initial therapy, assessed up to 3 years; margins of resection positive for tumor will not be considered disease recurrence).
Time Frame: Time from surgery to death or clinically apparent, biopsy confirmed recurrent or progressive disease after the completion of initial therapy, assessed up to 3 years; margins of resection positive for tumor will not be considered disease recurrence
Measure: Number; unit: DFS Probability
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 26
DFS Probability
  1-year disease free survival probability | 0.721
  2-year disease free survival probability | 0.641
  3-year disease free survival probability | 0.620

6. Secondary Outcome: Overall Survival
Description: Estimate overall survival (OS) in patients receiving the IRX-2 regimen. IRX-2 is currently being studied in an on-going Phase 2b clinical trial in patients with newly diagnosed Stage II, III, and IVA squamous cell carcinoma of the oral cavity (INSPIRE)
Time Frame: Time from surgery to death or confirmed recurrent or progressive disease, assessed up to 3 years
Measure: Number; unit: percentage of subjects
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 26
percentage of subjects
  First Year (%) | 92
  Second Year (%) | 73
  Third Year (%) | 69

7. Secondary Outcome: Number of Participants With High Lymphocyte Infiltration (LI) According to the Visual Analog Scale (VAS)
Description: Immunologic response features were extracted and quantified using a VAS of 0-100 mm to provide for a more continuous variable than the 0-4+ scale that is often used to assess histological responses. The scoring was such that 100 represented the maximum for any sample and 0 represented the lack of any parameter of interest.
  See publication of Berinstein, et al., 2012 for complete details.
Time Frame: On approximately Day 21 (last day of treatment) prior to undergoing post-treatment surgery
Population: Number of patients with high lymphocyte infiltration (LI).
Measure: Number; unit: participants with high LI (>34 mm) VAS
Arm/Group | IRX-2 Regimen
Number analyzed (Participants) | 25
participants with high LI (>34 mm) VAS | 18

8. Secondary Outcome: Relationship Between Overall Survival (OS) and Immune Competence (Lymphocyte Infiltration, LI) in Participants With High LI and Low LI
Description: After participants completed the IRX-2 regimen and the tumor resection was performed, tumor pathology was evaluated from tissue specimens obtained at tumor resection. Formalin-fixed, paraffin-embedded blocks, or unstained slides from the primary tumor were submitted to an independent pathology laboratory for hematoxylin and eosin staining, and evaluation of lymphocyte infiltration (LI). Participants were grouped into a "low LI" and "high LI" group based on the change in lymphocyte infiltration from the pretreatment tumor biopsy to the post-treatment tumor surgical resection. 5-year overall survival probabilities were then estimated (Kaplan-Meier) between the "low LI" and "high LI" groups
Time Frame: At time of surgery, after treatment with IRX-2 Regimen, assessed up to 5 years
Measure: Number; unit: 5-Year OS Probability
Groups:
- High Lymphocyte Infiltration (LI): Participants with high lymphocyte infiltration after treatment with the IRX-2 regimen
- Low Lymphocyte Infiltration: Participants with low lymphocyte infiltration after treatment with the IRX-2 regimen
Arm/Group | High Lymphocyte Infiltration (LI) | Low Lymphocyte Infiltration
Number analyzed (Participants) | 13 | 12
5-Year OS Probability | 0.80 | 0.50

ADVERSE EVENTS:
Time Frame: Primarily from the administration of cyclophosphamide to the time of surgery, except for Serious Adverse Events (reported up to 30 days after last dose of study medication)
Arm/Group | IRX-2 Regimen
All-Cause Mortality (participants affected / at risk) | 10/27
Serious Adverse Events (participants affected / at risk) | 7/27
Other Adverse Events (participants affected / at risk) | 23/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IRX-2 Regimen (N=27)
ASPIRATION PNEUMONIA (Infections and infestations) | 3 (3)
RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Respiratory Infection with Asthma
NECK ABSCESS (Infections and infestations) | 1 (1)
POSTOPERATIVE INFECTION (Infections and infestations) | 1 (1)
ALCOHOL WITHDRAWAL (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IRX-2 Regimen (N=27)
CONSTIPATION (Gastrointestinal disorders) | 4 (4)
DIZZINESS (General disorders) | 4 (4)
FATIGUE (General disorders) | 3 (3)
HEADACHE (General disorders) | 8 (8)
INJECTION SITE PAIN (General disorders) | 6 (6)
NAUSEA (General disorders) | 6 (6)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3)
INJECTION SITE DISCOMFORT (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less